CLINICAL TRIAL: NCT04101474
Title: Role Of Ketamine in Treatment-Resistant Major Depressive Disorder And Its Effect on Suicidality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, G.A. Khedr, Role Of Ketamine in treatment-Resistant Major Depressive Disorder And its Effect on Suicidality., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ketamine with TRD
Record Dates: First submitted 2019-09-22; First posted 2019-09-24 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The Sequentially Numbered, Opaque, Sealed Envelope technique (Schulz and Grimes, 2002) was employed: the randomization group was listed on paper and preserved in an opaque sealed envelope with a serial number. When a patient agreed to participate, the pharmacy (care provider) opened the sealed envelope and assigned the patient to the appropriate treatment group on the morning of their first infusion.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine group (Active Comparator): This group had ketamine
  Interventions: Drug: Ketamine
- Placebo group (No Intervention): This group had not take ketamine

INTERVENTIONS:
Drug: Ketamine — Ketamine is a high-affinity, noncompetitive N-methyl-D- aspartate (NMDA) glutamate receptor antagonist it has been used in anesthesiology for more than 50 years the time course of antidepressant response to ketamine is characterized by an initial reduction in depressive symptoms within 2 h
  Arms: Ketamine group

SUMMARY:
In this study we will assess the effect of Ketamine infusion on depressive symptoms and in particular its effect on Suicidal behavior, ideation and thoughts in patients with treatment- resistant MDD.

DETAILED DESCRIPTION:
A Twice repetition of IV infusion of 0.5 mg/kg of ketamine produces an antidepressant response in individuals with treatment-resistant MDD

The work aims to:

1. To assess the onset of action and degree of improvement and the duration of antidepressant effect of ketamine in a sample of patients with treatment -resistant major depressive disorder.
2. To find out whether the onset of Ketamine antidepressant effect is associated with an improvement of suicidality in those patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients fulfilling diagnostic criteria of treatment-resistant MDD.
2. Presence of suicidal risk.
3. No comorbid medical or neurological conditions.
4. Age above 18 years old.
5. Both gender.
6. Informed written consent from the patient or his legitimate.

Exclusion Criteria:

1. Presence of perceptual disturbance.
2. History of sensitivity to ketamine.
3. Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Role of Ketamine as Antidepressant | 1 year
  the onset of action and degree of improvement and the duration of antidepressant effect of ketamine in a sample of patients with treatment -resistant major depressive disorder.
Effect of Ketamine on Suicidality | 1 year
  finding out whether the onset of Ketamine antidepressant effect is associated with an improvement of suicidality in those patients

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt